CLINICAL TRIAL: NCT02585674
Title: A 21-Week, Open-label, Randomized, Controlled, Parallel-group, Multi-center Study Evaluating the Efficacy and Safety of HOE901-U300 Administered According to a Device-Supported Treat-to-target Regimen Versus Routine Titration in Patients With Type 2 Diabetes Mellitus
Brief Title: Comparison of MyStar DoseCoach to Routine Titration in Adult Patients With Type 2 Diabetes Mellitus Using Toujeo
Acronym: AUTOMATIX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC13470; 2014-004533-13 (EudraCT Number); U1111-1165-9001 (Other: UTN)
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MyStar DoseCoach (Experimental): MyStar DoseCoach - Device-supported treat-to-target regimen. Insulin glargine is administered subcutaneously on top of potential background therapy using oral anti-diabetic drug(s) or GLP1 RA injectable antihyperglycemic drug(s).
  Interventions: Drug: Insulin glargine (U300); Device: MyStar DoseCoach
- Routine Titration (Active Comparator): Routine Titration - Routine titration defined by the Investigator. Insulin glargine is administered subcutaneously on top of potential background therapy using oral anti-diabetic drug(s) or GLP1 RA injectable antihyperglycemic drug(s).
  Interventions: Drug: Insulin glargine (U300)

INTERVENTIONS:
Drug: Insulin glargine (U300) — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: HOE901
Device: MyStar DoseCoach — Glucose meter
  Arms: MyStar DoseCoach

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of the MyStar DoseCoach (Long-acting Insulin Glargine Titration Meter) device-supported treat-to-target regimen relative to a routine titration regimen in the percentage of patients reaching glycemic target, ie, with a mean fasting self-monitored plasma glucose (FSMPG) value within the target range of 90-130 mg/dL (5.0-7.2 mmol/L) without a severe hypoglycemic episode during the 16-week on-treatment period.

Secondary Objective:

To assess the efficacy, safety, and adherence/satisfaction of MyStar DoseCoach

DETAILED DESCRIPTION:
The maximum study duration will be 21 weeks per patient that will consist of a 4-week screening period, a 16-week treatment period, and 1-week follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Patients with type 2 diabetes mellitus diagnosed at least one year before the screening visit.
* Patients who are insulin naïve (and considered by the investigator to be appropriate candidates for basal insulin therapy), or treated with basal insulin as their only insulin.
* HbA1c between 7.5% and 11% (inclusive) at screening.
* Fasting SMPG >130 mg/dL at first screening and FSMPG >130 mg/dL at randomization.
* Signed informed consent.

Exclusion criteria:

* Aged <18 years.
* Diabetes other than type 2 diabetes mellitus.
* MyStar DoseCoach device is not appropriate for the patient or use of device is otherwise contraindicated (in the opinion of the Investigator).
* Conditions/situations that are contraindications or off-label use according to Summary of Product Characteristics (SmPCs) of Oral Anti-Diabetes Drugs (OADs) and/or GLP-1 receptor agonists when applicable (prescribed), or insulin glargine and as defined in the national product label.
* Patients not on stable dose of glucose lowering therapy including OADs, GLP-1 receptor agonists, or basal insulin therapy, for the last 3 months (stable basal insulin therapy defined as maximum change in insulin dose of +/- 20%).
* Patients using mealtime insulin (short acting analogue, human regular insulin, or premix insulin) for more than 10 days in the last 3 months before screening visit.
* Patients with hypoglycemia unawareness.
* Patients with severe hypoglycemia in the past 90 days.
* Hospitalization in the past 30 days.
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for one week or more within 90 days prior to the time of screening.
* Unable to meet specific protocol requirements (eg, inability to perform blood glucose measurements, manage their own insulin glargine administration, or deemed unlikely to safely manage titration based on guidance by their health care provider or HCP, etc.), because of a medical condition or because the patient is under legal guardianship.
* Patients with cognitive disorders, dementia, or any neurologic disorder that would affect a patient's ability to participate in the study, including the inability to understand study requirements or to give complete information about adverse symptoms.
* Conditions/situations such as:
* Patients with conditions/concomitant diseases precluding their safe participation in this study (eg, active malignant tumor, major systemic diseases, presence of clinically significant diabetic retinopathy or presence of macular edema likely to require treatment within the study period, etc.),
* Patients unable to fully understand study documents and to complete them. Patients who have a caregiver together with whom they can fulfill all study requirements are eligible,
* Patient is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Within the last 3 months prior to screening: history of myocardial infarction, unstable angina, acute coronary syndrome, revascularization procedure, or stroke requiring hospitalization.
* Severe or uncontrolled Congestive Heart Failure (New York Heart Association [NYHA] functional classification III and IV); or inadequately controlled hypertension at the time of screening with a resting systolic or diastolic blood pressure >180 mmHg or >95 mmHg, respectively.
* Pregnant or breast-feeding women or women who intend to become pregnant during the study period as glycemic control may be unstable and insulin doses may be variable during this period.
* Women of childbearing potential (premenopausal, not surgically sterile for at least 3 months prior to the time of screening) must use an effective contraceptive method throughout the study. Effective methods of contraception include barrier methods (in conjunction with spermicide), hormonal contraception, or use of an intrauterine device (IUD) or intrauterine hormone-releasing system (IUS).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching fasting SMPG target range 90-130 mg/dL (5.0-7.2 mmol/L) at Week 16 (mean of the last 5 readings recorded over the last 2 weeks) without a severe hypoglycemic episode during the 16-week on-treatment period | Baseline to Week 16

SECONDARY OUTCOMES:
Percentage of patients reaching fasting SMPG target range of 90-130 mg/dL (5.0-7.2 mmol/L), (mean of the last 5 readings recorded over the last 2 weeks) without severe and/or confirmed hypoglycemic events | Baseline to Week 16
Percentage of patients reaching laboratory FPG target range (90-130 mg/dL) without severe hypoglycemia | Baseline to Week 16
Mean FSMPG glucose change from baseline (mean of the last 5 readings recorded over the last 2 weeks) | Baseline to Week 16
Time to reach the first fasting SMPG target range of 90-130 mg/dL (5.0-7.2 mmol/L) | Baseline to Week 16
Mean FPG glucose change from baseline | Baseline to Week 16
Mean HbA1c change from baseline | Baseline to Week 16
Percentage of patients reaching HbA1c of <7.5% and <7% | Week 16
Percentage of patients with hypoglycemic events | Baseline to Week 16
Number of hypoglycemic events | Baseline to Week 16
Percentage of patients with adverse events | Baseline to Week 16
Percentage of patients with serious adverse events | Baseline to Week 16
Assessment of satisfaction with diabetes treatment using Diabetes Treatment Satisfaction Questionnaire | Baseline to Week 16
Assessment of fear of hypoglycemia using Hypoglycemia Fear Survey-II | Baseline to Week 16
Assessment of emotional well-being using WHO-5 well-being index | Baseline to Week 16
Assessment of diabetes-related emotional stress using Diabetes Distress Scale | Baseline to Week 16
Assessment of satisfaction with glucose monitoring using the Glucose Monitoring Satisfaction Survey | Baseline to Week 16
Assessment of device Ease of Use using Ease of Use questionnaire | Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (19):
- Germany (9):
  - Investigational Site Number 276002, Berlin
  - Investigational Site Number 276001, Dresden
  - Investigational Site Number 276007, Essen
  - Investigational Site Number 276003, Heidelberg
  - Investigational Site Number 276010, Künzing
  - Investigational Site Number 276005, Neumünster
  - Investigational Site Number 276004, Oldenburg in Holstein
  - Investigational Site Number 276006, Pirna
  - Investigational Site Number 276008, Sulzbach-Rosenberg
- United Kingdom (10):
  - Investigational Site Number 826003, Airdrie
  - Investigational Site Number 826002, Belfast
  - Investigational Site Number 826011, Bristol
  - Investigational Site Number 826001, Chester
  - Investigational Site Number 826006, Dumfries
  - Investigational Site Number 826008, East Kilbride
  - Investigational Site Number 826005, Larbert
  - Investigational Site Number 826010, Londonderry
  - Investigational Site Number 826009, Swansea
  - Investigational Site Number 826007, Taunton

REFERENCES:
- [Derived] Ritzel R, Harris SB, Baron H, Florez H, Roussel R, Espinasse M, Muehlen-Bartmer I, Zhang N, Bertolini M, Brulle-Wohlhueter C, Munshi M, Bolli GB. A Randomized Controlled Trial Comparing Efficacy and Safety of Insulin Glargine 300 Units/mL Versus 100 Units/mL in Older People With Type 2 Diabetes: Results From the SENIOR Study. Diabetes Care. 2018 Aug;41(8):1672-1680. doi: 10.2337/dc18-0168. Epub 2018 Jun 12. PMID 29895556